CLINICAL TRIAL: NCT01663272
Title: A Trial of Cabozantinib (XL184) and Gemcitabine in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.105; HUM 62927 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-07-24; First posted 2012-08-13 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Cancer
Keywords: oncology; pancrease
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — cabozantinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cabozantinib with gemcitabine (Experimental): The Study Treatment Period will consist of continued treatment during which time patients will receive cabozantinib and gemcitabine until either disease progression or the occurrence of unacceptable drug-related toxicity
  Interventions: Drug: CABOZANTINIB; Drug: gemcitabine

INTERVENTIONS:
Drug: CABOZANTINIB — Daily oral cabozantinib administered days -7 until disease progression, intolerable adverse event(s) or patient choice.
  Other Names: XL184
Drug: gemcitabine — Gemcitabine administered intravenously on days 1, 8, and 15 every 28 days.
  Other Names: Gemzar

SUMMARY:
Gemcitabine is considered one of the standard drugs for advanced pancreatic cancer and is approved by the FDA to treat it. Cabozantinib is a new drug that has demonstrated effectiveness against pancreatic cancer in laboratory experiments, especially when given with gemcitabine. Initial studies with cabozantinib in pancreatic cancer have shown some activity against the disease. The purpose of this study is to determine the safest and highest dose of cabozantinib that can be given together with standard doses of gemcitabine in patients with pancreatic cancer. This study will determine the safety and tolerability of this two drug combination.

DETAILED DESCRIPTION:
Preclinical work at the University of Michigan has demonstrated that inhibition of c-Met with cabozantinib prevented the development of metastatic disease in an intra-cardiac injection model in NOD/SCID mice. Additionally, the combination of cabozantinib and gemcitabine demonstrated improved tumor control compared to either agent alone in a relevant orthotopic implantation mouse model.

Combining gemcitabine with the c-Met inhibitor cabozantinib in advanced pancreatic cancer is a novel strategy that takes advantage of an established cytotoxic agent with one that targets a pathway known to be important for the growth, dissemination, and resistance of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed pancreatic carcinoma.
2. locally advanced unresectable disease, metastatic disease, or recurrent disease following surgical therapy.
3. ≥ 18 years old.
4. Life expectancy of greater than 12 weeks.
5. ECOG performance status ≤1 (Karnofsky ≥70%) (See Appendix A).
6. adequate organ and marrow function as follows:
7. capable of understanding and complying with the protocol requirements and has signed the informed consent document.
8. use medically accepted barrier methods of contraception
9. women of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

1. neuroendocrine tumors of the pancreas.
2. more than 1 prior systemic treatment regimen for pancreatic cancer. may have received prior neoadjuvant or adjuvant therapy, including gemcitabine, provided 6 months have elapsed from completion of that treatment and the start of study therapy.
3. Previous gemcitabine therapy for advanced pancreatic cancer. Patients who have had chemotherapy within 4 weeks, nitrosoureas/mitomycin C within 6 weeks, or monoclonal antibody within 6 weeks prior to planned initiation of study treatment.
4. prior treatment with a small molecule kinase inhibitor or a hormonal therapy within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment.
5. have received an investigational agent within 28 days of the first dose of study treatment or 5 half-lives of the compound or active metabolite, whichever is longer.
6. have received radiation therapy within 14 days of study treatment.
7. have not recovered from toxicity due to all prior therapies (i.e., return to pretherapy baseline or to CTCAE Grade 0 or 1) except alopecia and non-clinically significant AEs.
8. known brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Zhen DB, Griffith KA, Ruch JM, Camphausen K, Savage JE, Kim EJ, Sahai V, Simeone DM, Zalupski MM. A phase I trial of cabozantinib and gemcitabine in advanced pancreatic cancer. Invest New Drugs. 2016 Dec;34(6):733-739. doi: 10.1007/s10637-016-0376-1. Epub 2016 Jul 21. PMID 27439894

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level -1: 20 mg of cabozantinib PO daily administered days -7 until disease progression, intolerable adverse event(s) or patient choice.
  800mg/m^2 of gemcitabine administered intravenously on days 1, 8, and 15 every 28 days.
- Dose Level 1: 20 mg of cabozantinib PO daily administered days -7 until disease progression, intolerable adverse event(s) or patient choice.
  1000mg/m^2 of gemcitabine administered intravenously on days 1, 8, and 15 every 28 days.
- Dose Level 2: 40 mg of cabozantinib PO daily administered days -7 until disease progression, intolerable adverse event(s) or patient choice.
  1000mg/m^2 of gemcitabine administered intravenously on days 1, 8, and 15 every 28 days.
Period: Overall Study
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2
Started | 5 | 6 | 1
Completed | 5 | 6 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cabozantinib With Gemcitabine: Patients received daily oral cabozantinib, at 20mg or 40mg, administered days -7 until disease progression, intolerable adverse event(s) or patient choice AND Gemcitabine at 800mg/m^2 or 1000mg/m^2 administered intravenously on days 1, 8, and 15 every 28 days.
Arm/Group | Cabozantinib With Gemcitabine
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 60.5 [41 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The MTD is defined at the highest dose level at which ≤25% of patients experience a dose-limiting toxicity (DLT).
Time Frame: 5 weeks
Measure: Number; unit: mg
Groups:
- Cabozantinib With Gemcitabine: The Study Treatment Period will consist of continued treatment during which time patients will receive cabozantinib and gemcitabine until either disease progression or the occurrence of unacceptable drug-related toxicity
  Cabozantinib: Daily oral cabozantinib (20mg OR 40mg) administered days -7 until disease progression, intolerable adverse event(s) or patient choice.
  Gemcitabine: Gemcitabine (800mg/m^2 OR 1000mg/m^2) administered intravenously on days 1, 8, and 15 every 28 days.
Arm/Group | Cabozantinib With Gemcitabine
Number analyzed (Participants) | 12
mg | NA — The MTD could not be determined as too many patients experienced toxicity at all dose levels.

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival (PFS, a secondary endpoint) will be calculated from day-7 of cycle 1 of study treatment, until documented disease progression or death. Patients removed from treatment for progression or other reasons will be followed for 30 days after their last dose.
Time Frame: day-7 of cycle 1 until 30 days post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib With Gemcitabine
Number analyzed (Participants) | 12
months | 4.7 [1.4 to 9.7]

ADVERSE EVENTS:
Groups:
- Cabozantinib With Gemcitabine: Adverse events were pooled for all treated patients and were not collected by dose level. Patients received daily oral cabozantinib, at 20mg or 40mg, administered days -7 until disease progression, intolerable adverse event(s) or patient choice AND Gemcitabine at 800mg/m^2 or 1000mg/m^2 administered intravenously on days 1, 8, and 15 every 28 days.
Arm/Group | Cabozantinib With Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib With Gemcitabine (N=12)
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 (1)
Death, NOS (General disorders) | 1 (1)
Flu Like Symptoms (Infections and infestations) | 1 (1)
Bile Duct Stenosis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib With Gemcitabine (N=12)
Anemia (Blood and lymphatic system disorders) | 5 (10)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 3 (3)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (11)
Fever (General disorders) | 3 (3)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (28)
Alkaline phosphatase increased (Investigations) | 7 (11)
Aspartate aminotransferase increased (Investigations) | 9 (16)
Blood bilirubin increased (Investigations) | 3 (8)
Creatinine increased (Investigations) | 2 (2)
Lipase increased (Investigations) | 1 (4)
Lymphocyte count decreased (Investigations) | 5 (9)
Neutrophil count decreased (Investigations) | 9 (21)
Platelet count decreased (Investigations) | 10 (24)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 10 (31)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The MTD could not be determined as too many patients experienced toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes